CLINICAL TRIAL: NCT01977950
Title: Nutritional Status and Care of Elderly People
Brief Title: Nutritional Risk and Nutritional Care Practices in the Hospitalized Elderly
Acronym: NUTRIELD
Status: Completed | Type: Observational
Sponsor: Oslo Metropolitan University (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Kari Almendingen, Professor, Oslo Metropolitan University
Other Study IDs: 1-2719007
Record Dates: First submitted 2013-10-31; First posted 2013-11-07 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Undernutrition; Malnutrition
Keywords: Undernutrition, Nutritional risk, NRS2002, nutritional care practices, hospital, elderly patients, nursing students
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to estimate the prevalence of nutritional risk and examine nutritional care practices in the hospitalized elderly at one large university hospital in Norway.

DETAILED DESCRIPTION:
A cross-sectional study was designed and carried out at a university hospital in Norway. The study was developed by a collegium at a nursing bachelor education program in a multidisciplinary collaboration with representatives from the university hospital and other experts. Data on nutritional risk and nutritional care practices of elderly patients were collected by 173 second year nursing students at the university college in question who were undergoing their acute and clinical care practice studies on 20 wards at the university hospital. Nine nutritional screening days were conducted in the academic years 2011/2012 and 2012/2013. On the screening days the students filled in the questionnaire for each patient, including questions about age, gender, length of hospital stay, normal weight in recent months, weight, height, BMI, nutritional risk and nutritional care practices. The students measured weight and height whenever possible, and screened the patients for nutritional risk. Data were collected by using a stratified sampling technique along with adequate power calculations to improve the representativeness of the sample. The researchers received anonymously completed questionnaires and screening forms from the students and never met the patients.

ELIGIBILITY:
Inclusion Criteria:

* All elderly (≥70 yrs) patients admitted on the included wards at 08.00 am on the screening days were asked to participate.

Exclusion Criteria:

* Terminal patients (assumed short-lived, <1 month), patients diagnosed with dementia and patients whom the ward staff found unfit to participate were excluded.

Min Age: 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients were recruited from a large University hospital in Norway. The university hospital covers about 10% of the Norwegian population, providing healthcare services for approximately half a million people living in urban and rural municipalities. The patient population is thus heterogenic with respect to ethnicity and socioeconomic factors. All somatic wards having nursing students in acute care clinical studies in autumn 2011 were included in the study. The study sample comprised 14 of 16 medical and surgical somatic wards. Additionally, one rehabilitation ward, one specialized short time unit, one emergency medicine ward, and one cardio-monitoring ward were included.
  Eligible patients were selected by the nursing students in cooperation with the ward nursing staff.
Sampling Method: Probability Sample
Enrollment: 508 (Actual)
Dates: Start 2011-09; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Nutritional risk | 9 screening days were conducted in 2011-2013
  Patients was screened for nutritional risk on 9 screening days conducted in the academic years of 2011/2012 and 2012/2103. The Nutritional Risk Screening Tool 2002 (NRS2002) was employed to identify nutritional risk in the patients.

SECONDARY OUTCOMES:
Nutritional care practices | 9 nutritional screening days were conducted in the period 2011-2013
  Questions regarding the nutritional care practices concerned weight measurements on admission and then weekly, conduction of nutritional risk screening, coding of undernutrition diagnosis (E43, E44, or E46) in line with the International Statistical Classification of Diseases and Related Health Problems (ICD-10), and initiation of nutritional measures.

CONTACTS AND LOCATIONS:
Overall Officials: Kari Almendingen, Professor, Study Chair — Oslo Metropolitan University